CLINICAL TRIAL: NCT01458197
Title: A Prospective, Multi-center, Placebo-controlled, Randomized, Double-blind, Phase 2 Study to Compare the Efficacy and Tolerability of Tarafenacin 0.2 mg and Tarafenacin 0.4 mg to Placebo Administered as Oral Daily Dose for Three Months in Patients Suffering From Overactive Bladder.
Brief Title: A Phase 2 Study to Compare the Efficacy and Tolerability of Tarafenacin 0.2 mg and Tarafenacin 0.4 mg to Placebo in Patients Suffering From Overactive Bladder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kwang Dong Pharmaceutical co., ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TFN-KD01
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Tarafenacin
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tarafenacin 0.2 mg (Experimental): Group 1
  Interventions: Drug: Tarafenacin 0.2 mg
- Tarafenacin 0.4 mg (Experimental): Group 2
  Interventions: Drug: Tarafenacin 0.4 mg
- Placebo (Placebo Comparator): Group 3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tarafenacin 0.2 mg — Capsule, qd, 12 weeks
  Arms: Tarafenacin 0.2 mg
Drug: Placebo — Capsule, qd, 12 weeks
  Arms: Placebo
Drug: Tarafenacin 0.4 mg — Capsule, qd, 12 weeks
  Arms: Tarafenacin 0.4 mg

SUMMARY:
1. Primary Objective:

   To evaluate the dose-response relationship of tarafenacin on efficacy.
2. Secondary Objectives:

   * To compare 12 weeks' efficacy of different doses of tarafenacin to that of placebo in patients suffering from Overactive Bladder. .
   * To compare the tolerability of different doses of tarafenacin to that of placebo in patients suffering from Overactive Bladder. .

ELIGIBILITY:
< Inclusion Criteria>

1. Patient of either sex aged 20 to 80 years (both inclusive);
2. Patients suffering from Overactive Bladder. based on cardinal symptoms (urgency, nocturia, frequency with or without urge incontinence) for at least 6 months prior to inclusion;
3. Patients who document the following symptoms in a 3-day diary card during the 14 day placebo run-in period

   * An average of ≥8 micturitions/24 hours;
   * Greater than or equal to three incontinence episodes
   * A total of ≥3 urgency episodes.

<Exclusion Criteria>

1. Patients with Clinically significant bladder outlet obstruction
2. Patients with predominant stress incontinence (>2 episode/week)
3. Patients with significant urogenital disease such as recurrent urinary tract infection (more than 2/6 months), bladder calculi, interstitial cystitis, urothelial tumours, hysterectomy or prostatectomy in the previous six months;
4. Females diagnosed with bladder cancer
5. Males diagnosed with bladder cancer
6. Patients with obstructive disease of the gastrointestinal tract, intestinal inflammatory disease, severe ulcerative colitis, inflammatory bowel disease, toxic megacolon, intestinal atony or paralytic ileum
7. Patients with acute Noehyeolgwangye disease, significant Cardiovascular Disease (arrhythmias, unstable angina pectoris, myocardial infarct, or are using a pacemaker), significant Orthostatic hypotension in the previous six months
8. Patients diagnosed with closed angle glaucoma or shallowness of the anterior chamber
9. Patients with any contraindication to antimuscarinic drugs

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
the change in the number of micturitions per 24 hours from baseline to the end of the 12 weeks treatment period | 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline to 12weeks in Number of urgency episodes | 12 weeks
Mean change from baseline to 12weeks in Number of incontinence episodes | 12 weeks
Mean change from baseline to 12weeks in Number of nocturia episodes | 12weeks
Mean change from baseline to 12weeks in Volume of urine passed per void | 12weeks
Mean change from baseline to 12weeks in score of King's Health Questionnaire | 12weeks

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea